CLINICAL TRIAL: NCT04185688
Title: The Reliability and Validity of the Functional Reach Test in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fatih Söke, Research Assistant, Gazi University
Other Study IDs: 2019-153
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Functional reach test; Reliability; Validity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Functional Reach Test: It measures the maximum distance an individual is able to reach forward beyond arm's length in the standing position when maintaining a fixed base of support.
  Biodex Balance System: Biodex Balance System is used to evaluate limits of stability. The limits of stability test consists of standing on the platform and leaning in eight directions to make a cursor displayed on the system's screen hit a target.
  Berg Balance Scale: It has 14 items, each of which is scored from 0 (i.e, severely impaired balance) to 4 (i.e., no balance impairment).
  Timed Up and Go test: It requires individual to stand up from an armed chair, walk 3m, turn around, walk back to the armed chair, and sit down again.
  Four square step test: It requires an individual to step over obstacles in various directions including forward, backward, and sideways.
  Interventions: Other: Functional Reach Test
- Healthy People: Functional Reach Test: It measures the maximum distance an individual is able to reach forward beyond arm's length in the standing position when maintaining a fixed base of support.
  Interventions: Other: Functional Reach Test

INTERVENTIONS:
Other: Functional Reach Test — The Functional Reach Test assesses balance by measuring the limits of stability while the patient reaches forwards as far as possible, having the arms in 90° flexion and without lifting the heels off the floor.

SUMMARY:
Loss of limits of stability ability is one of the major components of balance dysfunction in MS. The functional reach test is quick and clinically available tool for assessing limits of stability but reliability and validity of this test has not yet been systematically examined in people with Multiple Sclerosis.The aim of the study is to investigate reliability and validity of the functional reach test in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
At baseline, the functional reach test, limits of stability test by using Biodex Balance System, Berg Balance Scale, four step square test, and timed up and go test was applied to the patients with Multiple Sclerosis. The functional reach test was repeated after seven days from the first application to evaluate its reliability.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years,
* neurologist-diagnosed Multiple Sclerosis,
* Expanded Disability Status Scale (EDSS) score < 7,
* able to walk 20 m with or without aids,
* no MS exacerbation within the last 2 months,
* use of stable medication in the last 2 months.

Exclusion Criteria:

* other neurologic disorder,
* pregnancy,
* orthopedic problems affecting gait and stance,
* visual, auditory, orientational problems that could affect study results,
* cardiovascular, pulmonary, and humoral disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis who apply to Gazi University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Functional Reach Test | 30 seconds
  Functional Reach Test is clinically used to assess limits of stability.

SECONDARY OUTCOMES:
Biodex Balance System | 2 minutes
  Biodex Balance System is used to assess limits of stability.
Berg Balance Scale | 10 minutes
  Berg Balance Scale is used to assess functional balance. Berg Balance Scale is a 14-item related to daily living activities that is scored between 0 and 4. The maximum score is 56 points and higher scores represent better balance.
Four Square Step Test | 20 seconds
  Four Square Step Test is used to assess dynamic balance.
Timed Up and Go Test | 15 seconds
  Timed Up and Go Test is used to assess functional mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Söke, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganesan M, Kanekar N, Aruin AS. Direction-specific impairments of limits of stability in individuals with multiple sclerosis. Ann Phys Rehabil Med. 2015 Jun;58(3):145-50. doi: 10.1016/j.rehab.2015.04.002. Epub 2015 May 8. PMID 25960358
- [Background] Cameron MH, Nilsagard Y. Balance, gait, and falls in multiple sclerosis. Handb Clin Neurol. 2018;159:237-250. doi: 10.1016/B978-0-444-63916-5.00015-X. PMID 30482317
- [Background] Martins EF, de Menezes LT, de Sousa PH, de Araujo Barbosa PH, Costa AS. Reliability of the Functional Reach Test and the influence of anthropometric characteristics on test results in subjects with hemiparesis. NeuroRehabilitation. 2012;31(2):161-9. doi: 10.3233/NRE-2012-0786. PMID 22951711
- [Background] Katz-Leurer M, Fisher I, Neeb M, Schwartz I, Carmeli E. Reliability and validity of the modified functional reach test at the sub-acute stage post-stroke. Disabil Rehabil. 2009;31(3):243-8. doi: 10.1080/09638280801927830. PMID 18608433
- [Background] Lynch SM, Leahy P, Barker SP. Reliability of measurements obtained with a modified functional reach test in subjects with spinal cord injury. Phys Ther. 1998 Feb;78(2):128-33. doi: 10.1093/ptj/78.2.128. PMID 9474105
- [Background] Duncan PW, Studenski S, Chandler J, Prescott B. Functional reach: predictive validity in a sample of elderly male veterans. J Gerontol. 1992 May;47(3):M93-8. doi: 10.1093/geronj/47.3.m93. PMID 1573190
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941